CLINICAL TRIAL: NCT04493164
Title: Phase II Investigator Sponsored Study of CPX-351 in Combination With Ivosidenib for Patients With IDH1 Mutated Acute Myeloid Leukemia or High-Risk MDS
Brief Title: CPX-351 and Ivosidenib for the Treatment of IDH1 Mutated Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0096; NCI-2020-05258 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0096 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia With Gene Mutations; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Myeloid, Acute | interventions — ivosidenib; CPX-351; Injections; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CPX-351, ivosidenib) (Experimental): INDUCTION: Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5, and ivosidenib PO QD on days 1-28. Patients who do not achieve complete remission may receive a second cycle of induction therapy in the absence of disease progression or unacceptable toxicity. Patients achieving complete remission proceed to consolidation.
  CONSOLIDATION: Patients receive CPX-351 IV over 90 minutes on days 1 and 3, and ivosidenib PO QD on days 1-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive ivosidenib PO QD for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients who are experiencing clinical benefit and who have not experienced excessive toxicity after completion of 2 years of maintenance may be eligible to continue therapy after discussion with the principal investigator.
  Interventions: Drug: Ivosidenib; Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Drug: Ivosidenib — Given PO
  Other Names: AG-120; Tibsovo
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos

SUMMARY:
This phase II trial investigates how well CPX-351 and ivosidenib work in treating patients with acute myeloid leukemia or high-risk myelodysplastic syndrome that has IDH1 mutation. The safety of this drug combination will also be studied. IDH1 is a type of genetic mutation (change). Chemotherapy drugs, such as CPX-351, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ivosidenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. The purpose of this trial is to learn if CPX-351 in combination with ivosidenib can help to control IDH1-mutated acute myeloid leukemia or high-risk myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (ORR) including CR, CRh, CRi, MLFS, and PR of the combination of CPX-351 and ivosidenib in IDH1-mutated patients with AML or high-risk MDS

SECONDARY OBJECTIVES:

I. To assess safety of CPX-351 in combination with ivosidenib. II. To determine time to event endpoints including duration of response (DOR), event free survival (EFS) and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. Evaluate minimal residual disease (MRD) using multiparameter flow cytometry, cytogenetics and molecular evaluation.

II. To evaluate molecular and cellular biomarkers that may be predictive of antitumor activity and/or resistance to treatment including evaluation of 2HG, IDH1 and other co-occurring mutations and VAF levels before, during and after treatment.

OUTLINE:

INDUCTION: Patients receive CPX-351 intravenously (IV) over 90 minutes on days 1, 3, and 5, and ivosidenib orally (PO) once daily (QD) on days 1-28. Patients who do not achieve complete remission may receive a second cycle of induction therapy in the absence of disease progression or unacceptable toxicity. Patients achieving complete remission proceed to consolidation.

CONSOLIDATION: Patients receive CPX-351 IV over 90 minutes on days 1 and 3, and ivosidenib PO QD on days 1-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive ivosidenib PO QD for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients who are experiencing clinical benefit and who have not experienced excessive toxicity after completion of 2 years of maintenance may be eligible to continue therapy after discussion with the principal investigator.

After completion of study treatment, patients are followed up at 30 days, then monthly for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* IDH1-R132 mutated disease status as assessed by local laboratory. 2HG-producing IDH1 variants outside of R132 (i.e. R100) may be eligible after discussion with the principal investigator (PI)
* Treatment naive or relapsed/refractory AML who are eligible for intensive chemotherapy. Patients with high-risk MDS or MPN (defined as International Prognostic Scoring System Revised [IPSS-R] score ≥ 4 or dynamic [D]-IPSS ≥ 3) may also be eligible after discussion with the PI
* Adequate hepatic function (direct bilirubin ≤ 2 x upper limit of normal (ULN), Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 3 x ULN unless deemed to be related to underlying leukemia
* Adequate renal function including creatinine clearance ≥ 30 ml/min based on the Cockcroft-Gault equation.
* Willing and able to provide informed consent
* In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 7 days for cytotoxic or non-cytotoxic (immunotherapy) agents.
* Male subjects must agree to refrain from unprotected sex and sperm donation from initial study drug administration until 90 days after the last dose of study drug

Exclusion Criteria:

* Patients who have previously received CPX-351.
* Patients with any concurrent uncontrolled clinically significant medical condition including infection, laboratory abnormality, or psychiatric illness, which could place the patient at unacceptable risk of study treatment.
* The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions (1) intrathecal chemotherapy for prophylactic use or for controlled CNS leukemia. (2) use of hydroxyurea, and/or cytarabine (1 or 2 doses; up to 2 g/m2) for patients with rapidly proliferative disease is allowed before the start of study therapy.
* Patients with active graft-versus-host-disease (GVHD) status post stem cell transplant (patients without active GVHD on chronic suppressive immunosuppression and/or phototherapy for chronic skin GVHD are permitted after discussion with the PI).
* Patients with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
* Patients with symptomatic congestive heart failure (NYHA Class III or IV), unstable angina, or an ejection fraction < 45%.
* Patients with prior anthracycline exposure of > 360 mg/m2 daunorubicin (or equivalent), or > 210 mg/m2 daunorubicin (or equivalent) in patients with prior mediastinal radiation.
* QTc interval using Fridericia's formula (QTcF) > 470 msec. A prolonged QTc interval in the setting of right bundle branch block is permitted after discussion with the PI.
* Nursing women, women of childbearing potential (WOCBP) with positive urine or serum pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception

  a. Appropriate highly effective method(s) of contraception include oral or injectable hormonal birth control, IUD, and double barrier methods (for example a condom in combination with a spermicide).
* Subjects with a known medical history of progressive multifocal leukoencephalopathy (PML).
* Subjects taking strong CYP3A4 inducers are excluded from the study unless they can be transferred to other medications within ≥ 5 half-lives prior to dosing
* Patients with a diagnosis of acute promyelocytic leukemia (APL).
* Unresolved toxicities > grade 1 from prior treatment including chemotherapy, targeted therapy, immunotherapy, experimental agents, radiation, or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 3 years
  Defined as complete remission (CR) + complete remission with hematologic recovery (CRh) + complete remission with incomplete blood count recovery (CRi) + morphologic leukemia-free state (MLFS) + and partial remission (PR). Will be assessed based on revised International Working Group (IWG) response criteria for acute myeloid leukemia (AML). Estimated along 95% confidence interval.

SECONDARY OUTCOMES:
Duration of response | Up to 3 years
  Defined as the number of days from the date of initial response (PR or better) to the date of first documented disease progression/relapse or death, whichever occurs first.
Event-free survival | Up to 3 years
  Defined as the number of days from the date of treatment initiation (i.e., cycle 1 days 1 [C1D1]) to the date of documented treatment failure, relapses from CR, or death from any cause, whichever occurs first, and will be calculated for all patients. Will be estimated using the method of Kaplan and Meier.
Overall survival | Up to 3 years
  Will be estimated using the method of Kaplan and Meier.
Incidence of adverse events | Up to 3 years
  The severity of the adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. The number and percent of subjects with treatment-emergent adverse events will be summarized according to intensity and drug relationship, and categorized by System Organ Class and preferred term by dose level/part.

OTHER OUTCOMES:
Minimal residual disease (MRD) status | Up to 3 years
  The association between cellular biomarker, MRD, etc. and antitumor activity will be compared using Wilcoxon's rank sum test or Fisher's exact test, as appropriate. MRD negative status and exploratory biomarkers will be summarized graphically and with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: http://www.mdanderson.org — http://www.mdanderson.org